CLINICAL TRIAL: NCT00808366
Title: A Randomized, Parallel-Group, Multicentre, Open-Labelled, Active-Controlled Study to Assess the Efficacy, Safety and Tolerability of RV4104A Ointment Versus Bifonazole-Urea Ointment for the Complete Removal of the Clinically Infected Nail Plate Area in Patients With Toenail Onychomycosis
Brief Title: Efficacy and Safety of RV4104A Ointment in Onychomycosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Anne-Marie Schmitt, MD, Pierre Fabre Dermo Cosmetique
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV4104A2007593
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Keratolytic Agents; Antifungal Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RV4104A ointment (Experimental)
  Interventions: Drug: Keratolytic/Antifungal
- bifonazole-urea ointment (Active Comparator)
  Interventions: Drug: Keratolytic/Antifungal

INTERVENTIONS:
Drug: Keratolytic/Antifungal — Intial treatment with RV4104A ointment for 3 weeks. Subsequent topical antifungal treatment with bifonazole cream for 8 weeks.
  Arms: RV4104A ointment
Drug: Keratolytic/Antifungal — Initial treatment with bifonazole-urea ointment for 3 weeks. Subsequent topical antifungal treatment with bifonazole cream for 8 weeks.
  Arms: bifonazole-urea ointment

SUMMARY:
The purpose of the study is to evaluate the efficacy of RV4104A ointment versus bifonazole-urea ointment for the complete removal of the clinically infected nail plate area in patients with toenail onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of distal-lateral or lateral subungual onychomycosis of one great toenail (the target nail)
* Target nail plate showing ≥ 12.5% of clinically infected area
* Patient must have at least 2 mm of the proximal end of the target nail free of infection
* Target nail infection due exclusively to a dermatophyte (from both positive direct microscopy examination and positive fungal culture as reported by the central mycological laboratory)

Exclusion Criteria:

* Patient with more than 2 affected toenails
* Patient with psoriasis, lichen planus or other abnormalities that could result in clinically abnormal toenail(s)
* Patient with moccasin-type tinea pedis
* Patient who has received systemic antifungal therapy or topical antifungal nail lacquer within 3 months or any other topical antifungal therapy applied to the feet or toenails within 2 months prior to screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-06 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Complete removal of the clinically infected target nail plate area after treating for 3 weeks assessed by a blinded imaging expert's panel on the basis of standardized photographs | D21

SECONDARY OUTCOMES:
Complete removal of the clinically infected target nail plate area after treating for 3 weeks assessed by the investigator on the basis of clinical evaluation | D21
Patient self-assessment | D21, D77, D105
Clinical cure | D77, D105
Mycological cure | D105
Complete cure of onychomycosis | D105
Local tolerability | D7, D21
Adverse Event reporting | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Carle PAUL, Professor, Principal Investigator — Hôpital Purpan, Toulouse - FRANCE
Locations (1):
- Hôpital Purpan, Toulouse, France